CLINICAL TRIAL: NCT02988323
Title: Cervicovestibular Rehabilitation and Aerobic Exercise in Children and Youth With Persistent Symptoms Following a Sport-related Concussion: A Randomized Controlled Trial.
Brief Title: Cervicovestibular Physiotherapy and Aerobic Exercise in Concussion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sport Injury Prevention Research Centre (Other)
Collaborators: University of Calgary (Other)
Responsible Party: Principal Investigator, KSchneider, Assistant Professor, Sport Injury Prevention Research Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Conc-PT-02
Record Dates: First submitted 2016-10-12; First posted 2016-12-09 (Estimated); Last update posted 2016-12-09 (Estimated); Status verified 2016-12

CONDITIONS: Concussion
Keywords: sport concussion; cervical spine; vestibular rehabilitation; exercise; rehabilitation; children; youth
MeSH Terms: conditions — Brain Concussion; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cervicovestibular Physio (CV PT) (Experimental): In addition to the standard protocol of rest followed by exertion, the CV PT group will participate in a combination of cervical spine and vestibular rehabilitation as per a standardized treatment algorithm based on individual assessment findings. This form of therapy combines treatment techniques for both the cervical spine and vestibular system that are commonly used in physiotherapy practice. Cervical spine treatments may include neuromotor retraining, sensorimotor retraining, manual therapy, soft tissue techniques, and range of motion exercises. Vestibular rehabilitation may include gaze stabilization, habituation, standing balance, dynamic balance and canalith repositioning maneouvers.
  Interventions: Other: Cervicovestibular Physio (CV PT)
- Low-Level Aerobic Exercise (LLAE) (Experimental): Participants will exercise at 60% maximum heart rate for 15 minutes. This heart rate will be calculated by taking 220-age (in years) and multiplying by 0.6 to determine the target heart rate while performing the low level aerobic exercise. Aerobic exercises may include treadmill, walking or stationary cycling. Exercise will be performed 5-6 times per week independently at home and monitored by their parents. Individuals will be taught how to monitor their heart rate. This protocol has previously been found to be feasible and of minimal risk to participants.
  Interventions: Other: Low-Level Aerobic Exercise (LLAE)
- Combination (LLAE and CV PT) (Other): The combination group will complete a protocol that includes both the cervicovestibular physiotherapy and LLAE interventions described above. As described above, the study participants will be seen once weekly by the study physiotherapist for CV PT and also complete a protocol of LLAE at home.
  Interventions: Other: Combination (LLAE and CV PT)

INTERVENTIONS:
Other: Cervicovestibular Physio (CV PT) — See description in CVPT arm
  Arms: Cervicovestibular Physio (CV PT)
Other: Low-Level Aerobic Exercise (LLAE) — See description in LLAE arm
  Arms: Low-Level Aerobic Exercise (LLAE)
Other: Combination (LLAE and CV PT) — See description in LLAE and CVPT arm
  Arms: Combination (LLAE and CV PT)

SUMMARY:
Sport concussions are among the most commonly occurring injuries in sport and recreation and pose significant public health implications for Canadians. Many individuals who sustain a concussion recover in the initial 7-10 days but up to 74% of youth and 31% of adults may suffer from persistent symptoms. Little research is currently available evaluating the effects of treatment for individuals who are slower to recover following sport-related concussion. An initial RCT identified a significant treatment effect in individuals with persistent symptoms of dizziness, neck pain and/or headaches following sport-related concussion when treated with a combination of cervical and vestibular physiotherapy compared to a typical protocol of rest followed by graded exertion (Schneider et al, 2014). Low level aerobic exercise in combination with sport specific training may also be of benefit to facilitate recovery in children and youth following concussion (Gagnon et al, 2009, 2016). Further evaluation of these treatments is required to better understand the effects of each treatment in isolation and in combination. This trial will have the ability to inform future multifaceted clinical trials as well as clinical practice. Ultimately, identification of optimal treatment paradigms will lead to a decrease in persistent symptoms and functional alterations in children and youth from this commonly occurring injury.

DETAILED DESCRIPTION:
Although awareness regarding sport-related concussion is growing, rehabilitative strategies for this commonly occuring injury have been a focus of very little research. With the exception of our pilot RCT, no RCTs to date have evaluated the efficacy of cervical spine physiotherapy in combination with vestibular rehabilitation in sport-related concussion. Current evidence has suggested positive effects of low-level aerobic exercise in youth and adults who are slow to recover following a concussion (Gagnon et al, 2016). However, low-level aerobic exercise has not yet been compared to cervicovestibular physiotherapy. A shift in clinical practice (to implement cervicovestibular physiotherapy or low level aerobic exercise) is occurring, but a direct comparison of the effects of low level aerobic exercise and multimodal physiotherapy treatment has not yet been conducted. A combination of these two forms of treatment may be more beneficial than either in isolation. Thus, the combination of physiotherapy and low level aerobic exercise treatment also requires evaluation. Identification of management strategies for individuals with persistent symptoms following concussion is urgently required to inform practice and optimize treatment strategies in this commonly occuring health problem.

OBJECTIVES:

Primary Research Question:

1. Does cervical and vestibular rehabilitation (CVPT) 1) result in a greater proportion of individuals medically cleared to return to sport (yes/no); 2) improve quality of life compared to a control group of low level aerobic exercise (LLAE) (following an 8-week intervention in individuals with persistent symptoms of dizziness, neck pain and/or headaches following concussion)?

Secondary Research Questions:

1. Does a combination of CVPT and LLAE 1) result in a greater proportion of individuals medically cleared to return to sport; 2) Improve quality of life compared to CVPT or LLAE alone (following an 8-week intervention in individuals with persistent symptoms of dizziness, neck pain and/or headaches following concussion)?

Exploratory Research Questions:

1. Does cervical and vestibular rehabilitation (CVPT) result in a greater proportion of individuals medically cleared to return to sport compared to a control group of low level aerobic exercise (LLAE) (following an 8-week intervention in individuals with persistent symptoms of dizziness, neck pain and/or headaches following concussion) when stratified by subgroups based on time since injury, previous history of concussion, sex and age?
2. Does a combination of CVPT and LLAE result in a greater proportion of individuals medically cleared to return to sport compared to CVPT or LLAE alone when stratified by subgroups based on time since injury, previous history of concussion, sex and age?
3. What clinical characteristics predict response to treatment?
4. What changes in symptoms and clinical measures of cervical and vestibular function occur with treatment?
5. What changes in measures of disability, self-efficacy, neuropsychological and psychosocial function occur with treatment?
6. What other factors may affect treatment outcome (i.e. medical clearance) and quality of life in youth with persisting symptoms following concussion?

METHODS:

The study design is a single blind randomized controlled trial (RCT). Participants will be recruited through the University of Calgary Acute Sport Concussion Clinic and through community sport medicine offices, family physicians and allied health in the City of Calgary and surrounding areas.

All participants will undergo an initial physiotherapy assessment at inclusion into the study. This assessment will be repeated at the time of medical clearance to return to sport (if less than 8 weeks) or at 8 weeks following initiation of treatment. Participants will be randomized into a cervicovestibular physiotherapy intervention (CVPT) group, a low level aerobic exercise group (LLAE), or a combination of cervicovestibular physiotherapy and low level aerobic exercise group (combination). All study participants will meet weekly (30 minute appointment) with a study physiotherapist for eight weeks (or until the time of medical clearance to return to sport if clearance occurs prior to 8 weeks). All groups will follow a protocol of graded exertion as per the 4th International Consensus Guidelines (Zurich 2012, McCrory et al, 2013).

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria:

  * Ages 10-18 years of age
  * Diagnosed by the study sport medicine physician with a sport related concussion as per the 4th International Consensus guidelines
  * Persistent symptoms of dizziness, neck pain and/or headaches (>10 days and less than one year post injury) reported on the Sport Concussion Assessment Tool 3 (SCAT3) at initial or follow-up visit to the study sport medicine physician
  * Clinical findings suggesting cervical spine and/or vestibular involvement (i.e. limitations in cervical range of motion, positive clinical tests suggesting cervicogenic headaches, altered patterns of neuromotor control, alterations on dynamic visual acuity, dynamic balance, motion sensitivity, positive test for BPPV, etc)

Exclusion Criteria:

* • Inability to participate in physical activity for a reason other than sport related concussion

  * Inability to communicate in English language
  * Neurodevelopmental delays
  * Other orthopaedic injury affecting ability to participate
  * Medication known to affect neural adaptation as they may alter the response to treatment

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 96 (Estimated)
Dates: Start 2016-12; Primary Completion 2018-03 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Medical Clearance to return to sport | 8 weeks
  The primary outcomes of interest will be: 1) Medical clearance to return to sport by 8-weeks (as per the 4th International Consensus Guidelines on Concussion in Sport). Medical clearance was selected because it is the most clinically relevant measure and will reflect not only symptom resolution but also functional improvement. We have chosen to further standardize this outcome as follows to minimize risk of bias:
  1. Asymptomatic a rest
  2. Able to complete all steps of the return to play protocol with no recurrence of symptoms
  3. Able to return to school full time without accommodations
  4. No other clinical findings suggesting an inability to return to play Some individuals may choose not to return to sport (i.e. retire) or to have coaching decisions influence their return to sport (i.e. may return prior to medical clearance). Therefore, medical clearance to return to sport (as opposed to actual return) is felt to most accurately reflect recovery.
Pediatric Quality of Life | Change from Initial assessment to 8 weeks
  Paediatric Quality of Life Inventory (Peds-QL): The Pediatric Quality of Life Scale (PedsQL) is a measure of quality of life that is specific to children and measures four health domains including: Physical, emotional, social and school functioning. It is a measure that has demonstrated reliability and validity in multiple disease types in children, including traumatic brain injury.

SECONDARY OUTCOMES:
Sport Multidimensional Perfectionism Scale-2 | Change from Initial assessment to 8 weeks
Connor-Davidson Resilience Scale | Change from Initial assessment to 8 weeks
K6 Scale | Change from Initial assessment to 8 weeks
  The K6 scale is a 6-item rating scale designed to assess psychological distress. It was developed with support from the U.S. government's National Center for Health Statistics for use in the redesigned U.S. National Health Interview Survey (NHIS). As described in more detail in Kessler et al. (2003), the scale was designed to be sensitive around the threshold for the clinically significant range of the distribution of nonspecific distress in an effort to maximize the ability to discriminate cases of serious mental illness (SMI) from non-cases.
Supplemental Questions (Mrazick) | Change from Initial assessment to 8 weeks
  Questions related to distress about injury at the time of injury, time of assessment and belief to make a full recovery rated on a 0-10 point scale
Self-efficacy questionnaire for children (Gagnon et al, 2009) | Change from Initial assessment to 8 weeks
Global Rating of Change | Change from Initial assessment to 8 weeks
Numeric Pain Rating Scale (Neck Pain) | Change from Initial assessment to 8 weeks
  Neck pain rating from 0-10
Numeric Pain Rating Scale (Headache) | Change from Initial assessment to 8 weeks
  Headache rating from 0-10
Numeric Dizziness Rating Scale | Change from Initial assessment to 8 weeks
  Dizziness rating from 0-10
Patient Specific Functional Scale (PSFS) | Change from Initial assessment to 8 weeks
Activities-specific Balance Confidence Scale | Change from Initial assessment to 8 weeks
Dizziness Handicap Inventory | Change from Initial assessment to 8 weeks
Sport Concussion Assessment Tool 3 | Change from Initial assessment to 8 weeks
Dynamic Visual Acuity | Change from Initial assessment to 8 weeks
  Clinical test of dynamic visual acuity using ETDRS
Balance Error Scoring System | Change from Initial assessment to 8 weeks
Functional Gait Assessment | Change from Initial assessment to 8 weeks
  10 item standardized test of dynamic balance
Head Thrust Test | Change from Initial assessment to 8 weeks
Motion Sensitivity Test | Change from Initial assessment to 8 weeks
Cervical Flexor Endurance | Change from Initial assessment to 8 weeks
  Standardized test of cervical flexor endurance measured in seconds
Cervical Flexion Rotation Test (CFRT) | Change from Initial assessment to 8 weeks
Palpation for Segmental Tenderness (PST) | Change from Initial assessment to 8 weeks
  As per Schneider et al 2014, palpation for segmental tenderness in cervical spine
Cervical Rotation Side Flexion Test | Change from Initial assessment to 8 weeks
Joint Position Error (JPE) | Change from Initial assessment to 8 weeks
Walk While Talking Test | Change from Initial assessment to 8 weeks
Vestibular/Ocular Motor Screen (VOMS) | Change from Initial assessment to 8 weeks
  As per Mucha et al, 2014
Manual Spinal Examination (MSE) | Change from Initial assessment to 8 weeks
  As per Schneider et al, 2014
Actigraphy | Change from Initial Assessment to 8 weeks
  Use of a waist worn activity monitor to validly measure the amount of physical activity that an individual performs throughout their day.

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Schneider, Principal Investigator — University of Calgary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McCrory P, Meeuwisse WH, Aubry M, Cantu RC, Dvorak J, Echemendia RJ, Engebretsen L, Johnston K, Kutcher JS, Raftery M, Sills A, Benson BW, Davis GA, Ellenbogen R, Guskiewicz KM, Herring SA, Iverson GL, Jordan BD, Kissick J, McCrea M, McIntosh AS, Maddocks D, Makdissi M, Purcell L, Putukian M, Schneider K, Tator CH, Turner M. Consensus statement on concussion in sport: the 4th International Conference on Concussion in Sport, Zurich, November 2012. J Athl Train. 2013 Jul-Aug;48(4):554-75. doi: 10.4085/1062-6050-48.4.05. No abstract available. PMID 23855364
- [Background] Gagnon I, Galli C, Friedman D, Grilli L, Iverson GL. Active rehabilitation for children who are slow to recover following sport-related concussion. Brain Inj. 2009 Nov;23(12):956-64. doi: 10.3109/02699050903373477. PMID 19831492
- [Background] Schneider KJ, Meeuwisse WH, Nettel-Aguirre A, Barlow K, Boyd L, Kang J, Emery CA. Cervicovestibular rehabilitation in sport-related concussion: a randomised controlled trial. Br J Sports Med. 2014 Sep;48(17):1294-8. doi: 10.1136/bjsports-2013-093267. Epub 2014 May 22. PMID 24855132
- [Background] Schneider KJ, Iverson GL, Emery CA, McCrory P, Herring SA, Meeuwisse WH. The effects of rest and treatment following sport-related concussion: a systematic review of the literature. Br J Sports Med. 2013 Apr;47(5):304-7. doi: 10.1136/bjsports-2013-092190. PMID 23479489
- [Background] Gagnon I, Grilli L, Friedman D, Iverson GL. A pilot study of active rehabilitation for adolescents who are slow to recover from sport-related concussion. Scand J Med Sci Sports. 2016 Mar;26(3):299-306. doi: 10.1111/sms.12441. Epub 2015 Mar 3. PMID 25735821